CLINICAL TRIAL: NCT06174909
Title: In Vivo Comparative Study Calcium Hydroxide and Triple Antibiotic Paste in Emergency Pain Reduction
Brief Title: In Vivo Comparative Study of Calcium Hydroxide and Triple Antibiotic Paste in Intracanal Medicament in Emergency Pain Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Ahsen amin, Principal investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2022
Record Dates: First submitted 2023-09-09; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide (Experimental): Calcium hydroxide has antimicrobial properties and tissue altering effect,used into root canals for the purpose of inhibiting coronal invasion of bacteria from the oral cavity".
  Interventions: Drug: Calcium Hydroxide
- Triple antibiotic Paste (Active Comparator): Triple antibiotic paste is combination of ciprofloxcin,metronidazole,and minocycline,used into root canals for the purpose of inhibiting coronal invasion of bacteria from the oral cavity".
  Interventions: Drug: Triple Antibiotic paste

INTERVENTIONS:
Drug: Calcium Hydroxide — After completion of canal and shaping ,canal was dried and CH was placed as an intracanal medicament. A total of 100 mg of CH powder was dispensed and mixed with one drop of pro-pylene glycol on a clean and dry glass slab to prepare a thick paste-like consistency. This paste was carried into the canal and access opening was restored temporarily with temporary cement
  Arms: Calcium Hydroxide
Drug: Triple Antibiotic paste — After completion of cleaning and shaping ,canal was dried and tripe antibiotic was placed as intracanal medicament.It was prepared by removing the coating and crushing of antibiotic ciprofloxacin500mg,metronidazole 400mg,, and clindamycin tablets separately using a mortar and pestle. It was prepared by removing the coating and crushing of antibiotic ciprofloxacin500mg,metronidazole 400mg,, and clindamycin tablets separately using a mortar and pestle. This paste was placed gently compacted into the canal and access opening was restored with temporary cement
  Arms: Triple antibiotic Paste

SUMMARY:
Interappointment pain is a universal concern for clinician and patients alike which remain a significant challenge for dentalprofessional.The purpose of this study was to evaluate the effects of calcium hydroxide, and triple antibiotic paste as intra-canal medicaments in emergency pain reduction in patients undergoing endodontic treatment .

DETAILED DESCRIPTION:
Before commencing treatment, the complete procedure was explained to the patients and consent was obtained. Local anesthesia was administered, and the tooth was isolated under rubber dam. Access cavity preparation was done, and canals were explored using endodontic explorer (DG-16,). Working length was determined with No. 15 K-files using apex locater and was confirmed with radiovisiography . Cleaning and shaping were along with copious irrigation using 3% NaOCl and 0.9% saline . Canals will be dried and one of the following two medicaments will be inserted into the canals in random sequences

Group 1 :Calcium Hydroxide:

CH was placed as an intracanal medicament. Atotal of 100 mg of CH powder was dispensed and mixed with one drop of pro-pylene glycol on a clean and dry glass slab to prepare a thick paste-like consistency. This paste was carried into the canal , and access opening was restored temporarily with temporary cement

Group 2: Triple antibiotic paste:

It was prepared by removing the coating and crushing of antibiotic ciprofloxacin500mg,metronidazole 400mg,, and clindamycin tablets separately using a mortar and pestle. The crushed powder was passed through a fine sieve to remove heavy filler particles and obtain a fine powder. The ciprofloxacin, metronidazole, and clindamycin powders thus obtained were weighed separately and mixed in a 1:3 proportions respectively,to obtain triple antiobiotic mixture.A total 100 mg of this Ta mixture was dispensed and mixed with one drop of propylene glycol to get a thick paste-like consistency. This paste was placed gently compacted into the canal , and access opening was restored with temporary cement Before dismissal ,no antiobiotics will be prescribed and the patients who had been taking antibiotics will be recorded.Patient will be requested to stop antibiotics.They will be requested to stop analgesic.The preoperative pain experienced on the previous night will be recorded using visual analogue scale.Patient will be then instructed to record the degree of pain experienced after 2nd day ,7th day and 15 day postoperatively

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who agree to particapte in study 2. Patient with age between 18 to 60 years 3. single rooted teeth with closed apices included in the study 4. Patient diagnosed with Necrosed tooth with acute apical periodontitis will be included in the study.

Exclusion Criteria:

* 1. Teeth with incomplete root formation. 2. Severe periodontal problem. 3. Vertical or horizontal root fractures were excluded from the study 4. Retreatment cases will not included in study. 5. Patients with systemic problems, for example, diabetes and autoimmune disease, and so on, will not be selected for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Immediately after the procedure
  Pain after root canal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Islamabad, Pakistan